CLINICAL TRIAL: NCT03829683
Title: Vitamin C Infusion for TReatment in Sepsis and Alcoholic Hepatitis
Acronym: CITRIS-AH
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Virginia Commonwealth University (Other)
Collaborators: National Institute on Alcohol Abuse and Alcoholism (NIAAA) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: HM20014364; U01AA026966 (NIH)
Record Dates: First submitted 2019-01-17; First posted 2019-02-04 (Actual); Results first posted 2023-03-21 (Actual); Last update posted 2023-08-28 (Actual); Status verified 2023-08

CONDITIONS: Alcoholic Hepatitis; Sepsis
MeSH Terms: conditions — Hepatitis, Alcoholic; Sepsis | interventions — Ascorbic Acid; Glucose; Water

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: Study drug will be double-blind with matching placebo. Vitamin C 200mg/kg/24hours or placebo (Dextrose 5% in water) will be given intravenously every 6 hours for up to 96 hours of treatment.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Vitamin C infusion (ascorbic acid) (Active Comparator): Vitamin C 200mg/kg/24hours administered in four doses per day (given every 6 hours)
  Interventions: Drug: Vitamin C; Drug: Dextrose 5% in water
- Placebo (Placebo Comparator): Dextrose 5% in water 50 milliliters (mL) administered intravenously every 6 hours
  Interventions: Drug: Dextrose 5% in water

INTERVENTIONS:
Drug: Vitamin C — 200mg/kg/24hours
  Other Names: ascorbic acid; AscA; Ascor
  Arms: Vitamin C infusion (ascorbic acid)
Drug: Dextrose 5% in water — 50mL intravenously every 6 hours
  Other Names: D5W

SUMMARY:
The purpose of this research study is to test the safety, tolerability, and effectiveness of Vitamin C (ascorbic acid) intravenous infusion when used to treat alcoholic hepatitis (inflammation of the liver from heavy alcohol use) and sepsis (life-threatening complication of an infection).

DETAILED DESCRIPTION:
Alcoholic hepatitis is inflammation of the liver due to alcohol consumption. It can cause one or more of the following symptoms such as jaundice (yellow discoloration of the eyes and skin), pain on the right side of the abdomen, and is accompanied by an enlarged liver. Sepsis is a life-threatening complication of an infection. As the body tries to fight an infection it sends chemicals into the bloodstream. These chemicals that are trying to fight the infection can cause inflammation. This inflammation can cause damage to many body systems and make them fail. Patients with alcoholic hepatitis and sepsis have low levels of Vitamin C in the bloodstream. Vitamin C has been shown to reduce inflammation and organ dysfunction in patients with severe infections.

The investigators do not yet know if Vitamin C will be effective in alcoholic hepatitis. Taking Vitamin C by mouth is not effective as a treatment in people with this condition so participants will receive the Vitamin C intravenously (IV). Participants will be randomly assigned to receive either Vitamin C or a placebo given through an IV every six hours for four days.

ELIGIBILITY:
Inclusion Criteria:

1. Alcoholic Hepatitis diagnosed by one of the following methods:

   1. liver biopsy
   2. clinical diagnosis based on history of alcohol use, presence of jaundice (yellowing of skin), blood tests indicating liver injury, and absence of other causes of liver injury (autoimmune disease, viral hepatitis, drug toxicity)
2. Suspected or proven infection
3. Presence of systemic inflammatory response to infection (fever, hypothermia (low temperature), tachycardia (fast heart rate), leukocytosis (high white blood cell count), leukopenia (low white blood cell count), high respiratory (breathing) rate, or need for mechanical ventilation (a machine to assist in breathing).
4. Presence of organ failure due to the body's response to infection indicated by any of the following:

   1. Hypotension (low blood pressure) or need for medications to raise blood pressure
   2. Arterial hypoxemia (low blood oxygen) or need for high flow of oxygen
   3. High lactate level (blood test indicating active response to infection)
   4. Low urine output despite administration of intravenous fluids
   5. Low platelet count (blood test)
   6. Coagulopathy (decreased blood clotting ability based on a blood test)
   7. High bilirubin (blood test)
   8. Mental status changes (confusion or delirium)
5. Absence of drugs present on urine or blood tests that indicate the possibility of liver damage or mental status changes from other causes

Exclusion Criteria:

1. Allergy to Vitamin C
2. Unable to provide consent
3. Age less than 18 years
4. No intravenous access (IV line) in a patient needing glucose (blood sugar) checks more than twice daily
5. Presence of diabetic ketoacidosis (a serious complication of diabetes)
6. Inability of patient, legally authorized representative and/or physician to commit to full medical support
7. Pregnancy or breast feeding
8. Life expectancy less than 24 hours
9. Active or history of kidney stone
10. History of chronic kidney disease
11. History of glucose-6-phosphate deficiency (a low blood protein that can cause red blood cells to break down)
12. Active cancer (except non-melanoma skin cancer)
13. Uncontrolled gastrointestinal bleeding
14. Other causes of liver injury such as viruses, autoimmune disease, drug toxicity
15. History of severe liver cirrhosis complications including variceal bleeding within the last 3 months, large ascites (fluid accumulation in the abdomen) or hepatocellular carcinoma (liver cancer)
16. History of organ transplantation
17. Initial AST or ALT (blood test indicating a liver problem)
18. Presence of acetaminophen or other drugs on urine or blood toxicology test
19. Non-English speaking
20. Prisoner or other ward of the state

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Actual)
Dates: Start 2019-04-16 (Actual); Primary Completion 2022-03-31 (Actual); Study Completion 2022-06-23 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Arun J Sanyal, MD, Principal Investigator — Virginia Commonwealth University
Locations (1):
- Virginia Commonwealth University, Richmond, Virginia, United States

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Vitamin C Infusion (Ascorbic Acid) | Placebo
Started | 10 | 10
Completed | 5 | 8
Not Completed | 5 | 2
Not completed — Lost to Follow-up | 1 | 0
Not completed — Physician Decision | 3 | 1
Not completed — Withdrawal by Subject | 0 | 1
Not completed — Discharge from hospital | 1 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Vitamin C Infusion (Ascorbic Acid) | Placebo | Total
Number analyzed (Participants) | 10 | 10 | 20
Age, Continuous [Mean (Standard Deviation); unit: years] | 40.1 (9.5) | 48.4 (14.9) | 46.9 (12.5)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 7 | 7 | 14
  Male | 3 | 3 | 6
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 1 | 0 | 1
  Not Hispanic or Latino | 9 | 10 | 19
  Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 1 | 1 | 2
  White | 8 | 9 | 17
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 1 | 0 | 1
Region of Enrollment [Number; unit: participants]
  United States | 10 | 10 | 20

OUTCOME MEASURES:

1. Primary Outcome: Change in Model for End Stage Liver Disease (MELD) Score
Description: Change in MELD score from Day 0 to Day 4. MELD score ranges from 6 (least sick) to 40 (most sick) based on blood tests which ranks the degree of sickness from liver disease. The lab tests used to determine the MELD score are creatinine, bilirubin, and international normalized ratio (INR).
Time Frame: Baseline and 96 hours
Population: Labs were not collected from 4 participants on day 4 so change in MELD score could not be calculated for those participants and they are omitted from the analysis.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Vitamin C Infusion (Ascorbic Acid) | Placebo
Number analyzed (Participants) | 8 | 8
score on a scale
  All patients | -0.13 (7.0) | -2.9 (3.3)
  Patients alive at 4 weeks: number analyzed (Participants) | 4 | 5
  Patients alive at 4 weeks | -2.3 (5.2) | -2.4 (1.3)

2. Secondary Outcome: Change in Chronic Liver Failure-Sequential Organ Failure Assessment (CLIF-SOFA) Score
Description: A number that ranges from 0 (least sick) to 24 (most sick) and ranks the degree of sickness from liver failure and several other organ systems in a critically ill person. The score is determined by evaluating a person's liver function, kidney function, nervous system (brain), coagulation (blood clotting), circulation (blood pressure), and respiratory status (breathing)
Time Frame: Baseline and 96 hours
Population: Data not recorded for all participants
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Vitamin C Infusion (Ascorbic Acid) | Placebo
Number analyzed (Participants) | 1 | 4
score on a scale
  Baseline: number analyzed (Participants) | 1 | 3
  Baseline | 14 (NA) — Only 1 participant in this arm | 15.33 (0.577)
  Day 4: number analyzed (Participants) | 0 | 4
  Day 4 |  | 12.75 (1.708)

3. Secondary Outcome: Change in Aspartate Aminotransferase (AST) Level
Description: Standard blood test used to determine the severity and nature of liver problems.
Time Frame: Baseline and 96 hours
Measure: Mean (Standard Deviation); unit: IU/L
Arm/Group | Vitamin C Infusion (Ascorbic Acid) | Placebo
Number analyzed (Participants) | 7 | 8
IU/L | 176.0 (466.28) | -16.5 (53.07)

4. Secondary Outcome: Change in Alanine Aminotransferase (ALT) Level
Description: Standard blood test used to determine the severity and nature of liver problems.
Time Frame: Baseline and 96 hours
Measure: Mean (Standard Deviation); unit: IU/L
Arm/Group | Vitamin C Infusion (Ascorbic Acid) | Placebo
Number analyzed (Participants) | 7 | 8
IU/L | 62.71 (155.26) | 1.00 (14.65)

5. Secondary Outcome: Change in Total Bilirubin
Description: Standard blood test used to determine the severity and nature of liver problems.
Time Frame: Baseline and 96 hours
Measure: Mean (Standard Deviation); unit: mg/dL
Arm/Group | Vitamin C Infusion (Ascorbic Acid) | Placebo
Number analyzed (Participants) | 7 | 8
mg/dL | -0.30 (5.69) | 0.45 (5.79)

6. Secondary Outcome: Change in Alkaline Phosphatase
Description: Standard blood test used to determine the severity and nature of liver problems.
Time Frame: Baseline and 96 hours
Measure: Mean (Standard Deviation); unit: U/L
Arm/Group | Vitamin C Infusion (Ascorbic Acid) | Placebo
Number analyzed (Participants) | 7 | 8
U/L | -5.71 (67.90) | -7.50 (52.86)

7. Secondary Outcome: Change in Albumin
Description: Standard blood test used to determine the severity and nature of liver problems.
Time Frame: Baseline and 96 hours
Measure: Mean (Standard Deviation); unit: g/dL
Arm/Group | Vitamin C Infusion (Ascorbic Acid) | Placebo
Number analyzed (Participants) | 7 | 8
g/dL | -0.10 (0.71) | 0.06 (0.99)

8. Secondary Outcome: Number of Treatment-related Adverse Events as Assessed by CTCAE v5.0
Description: Observation about the need to change the dose of study medication and symptoms such as headache, dizziness, dry mouth, nausea, vomiting, flushing, rash, or hypotension (low blood pressure)
Time Frame: up to 96 hours
Measure: Number; unit: Adverse Events
Arm/Group | Vitamin C Infusion (Ascorbic Acid) | Placebo
Number analyzed (Participants) | 10 | 10
Adverse Events | 12 | 11

9. Secondary Outcome: Changes to Corrected QT Interval (QTc)
Description: An electrocardiogram (ECG or test of the electrical activity of the heart) is performed to determine if there are changes to the heart rhythm.
Time Frame: Baseline and 96 hours
Measure: Mean (Standard Deviation); unit: milliseconds
Arm/Group | Vitamin C Infusion (Ascorbic Acid) | Placebo
Number analyzed (Participants) | 6 | 6
milliseconds | -10.00 (29.47) | -58.17 (88.56)

10. Secondary Outcome: Changes to Urine pH
Description: Urine samples are collected to determine changes in pH (acidity) that could indicate a risk for kidney stones. The pH scale ranges from 0 to 14, with smaller numbers meaning more acidic and higher numbers meaning more basic. A pH of 7 is considered to be neutral. Normal levels of urine pH range from 4.6 - 8 on the pH scale.
Time Frame: Baseline and 96 hours
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Vitamin C Infusion (Ascorbic Acid) | Placebo
Number analyzed (Participants) | 6 | 6
units on a scale | 5.31 (2.01) | 5.17 (0.41)

11. Secondary Outcome: Changes to Urine Microscopy
Description: Urine samples are collected to check for the presence of crystalluria (microscopic crystals) that could indicate a risk for kidney stones.
Time Frame: Baseline and 96 hours
Measure: Count of Participants; unit: Participants
Arm/Group | Vitamin C Infusion (Ascorbic Acid) | Placebo
Number analyzed (Participants) | 8 | 6
Participants
  Number of participants with crystalluria at baseline | 0 | 0
  Number of patients with crystalluria at Day 4 | 0 | 0

12. Secondary Outcome: Changes to Level of Medical Care
Description: Documentation of the need for more intensive medical care such as ventilator (breathing machine) or vasopressors (intravenous medications use increase blood pressure) when not needed at baseline
Time Frame: up to 168 hours
Measure: Count of Participants; unit: Participants
Arm/Group | Vitamin C Infusion (Ascorbic Acid) | Placebo
Number analyzed (Participants) | 10 | 10
Participants | 2 | 1

13. Secondary Outcome: ICU-free Days
Description: The number of days not spent in an intensive care unit (ICU)
Time Frame: Day 28
Measure: Mean (Standard Deviation); unit: days
Arm/Group | Vitamin C Infusion (Ascorbic Acid) | Placebo
Number analyzed (Participants) | 10 | 10
days | 16.40 (14.17) | 13.20 (13.06)

14. Secondary Outcome: Number of Deaths Due to Any Cause
Description: Any cause of death that is anticipated or unanticipated
Time Frame: Day 28
Measure: Number; unit: Deaths
Arm/Group | Vitamin C Infusion (Ascorbic Acid) | Placebo
Number analyzed (Participants) | 10 | 10
Deaths | 4 | 3

15. Secondary Outcome: Number of Deaths Due to Any Cause
Description: Any cause of death that is anticipated or unanticipated
Time Frame: Day 90
Measure: Number; unit: Deaths
Arm/Group | Vitamin C Infusion (Ascorbic Acid) | Placebo
Number analyzed (Participants) | 10 | 10
Deaths | 5 | 4

16. Secondary Outcome: Hospital-free Days
Description: The number of days spent outside of the hospital
Time Frame: Day 90
Measure: Mean (Standard Deviation); unit: days
Arm/Group | Vitamin C Infusion (Ascorbic Acid) | Placebo
Number analyzed (Participants) | 5 | 8
days | 58.40 (32.91) | 48.88 (33.04)

ADVERSE EVENTS:
Time Frame: Up to 90 days after drug infusion
Arm/Group | Vitamin C Infusion (Ascorbic Acid) | Placebo
All-Cause Mortality (participants affected / at risk) | 5/10 | 4/10
Serious Adverse Events (participants affected / at risk) | 2/10 | 0/10
Other Adverse Events (participants affected / at risk) | 7/10 | 5/10
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Vitamin C Infusion (Ascorbic Acid) (N=10) | Placebo (N=10)
Weakness, hospitalization (General disorders) | 1 (1) | 0 (0)
Acute kidney injury (Renal and urinary disorders) | 1 (1) | NA
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Vitamin C Infusion (Ascorbic Acid) (N=10) | Placebo (N=10)
Hypokalemia (Metabolism and nutrition disorders) | 1 (1) | 3 (3)
Abdominal pain (Gastrointestinal disorders) | 1 (1) | 0 (0)
Bladder spasm (Renal and urinary disorders) | 0 (0) | 1 (1)
Deep vein thrombosis (Vascular disorders) | 1 (1) | 0 (0)
Electrocardiogram QT corrected interval (Investigations) | 1 (1) | 0 (0)
Hyperglycemia (Metabolism and nutrition disorders) | 1 (1) | 2 (2)
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Hypomagnesemia (Metabolism and nutrition disorders) | 1 (1) | 0 (0)
Hypophospahtemia (Metabolism and nutrition disorders) | 1 (1) | 4 (4)
Hypotension (Cardiac disorders) | 0 (0) | 1 (1)
QT interval prolonged (Investigations) | 1 (1) | 0 (0)
Vomiting (Gastrointestinal disorders) | 1 (1) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2020-01-21): https://cdn.clinicaltrials.gov/large-docs/83/NCT03829683/Prot_SAP_001.pdf
  • Informed Consent Form (2018-12-20): https://cdn.clinicaltrials.gov/large-docs/83/NCT03829683/ICF_000.pdf